CLINICAL TRIAL: NCT00762489
Title: Comparison of Temporal Artery, Axillary, and Rectal Temperatures in Newborn Patients in the Well Baby Nursery.
Brief Title: Comparison of Three Methods of Taking Temperatures in the Well Baby Nursery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Michael F. Bruno, MD, Christiana Care Health Systems
Allocation: Non-Randomized | Model: Single Group
Other Study IDs: 28148
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-04

CONDITIONS: Newborn Infants
Keywords: Temporal artery thermometry; Rectal temperature; Axillary temperature; Newborns; Temperature measurement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAT vs. RT (Other): This arm is comparing the Temporal Artery Thermometer (TAT) temperature to the Rectal Temperature (RT).
  Interventions: Other: Temporal artery thermometer temperature
- TAT vs. AT (Other): This arm is comparing the Temporal Artery Thermometer (TAT) temperature to the Axillary Temperature (AT).
  Interventions: Other: Temporal artery thermometer temperature

INTERVENTIONS:
Other: Temporal artery thermometer temperature — Newborn infants had a temporal artery temperature taken within a few minutes of the axillary and rectal temperatures. The axillary and rectal temperatures are taken via methods which are standard of care.
  Other Names: Exergen TAT-5000 TemporalScanner Exergen Corp; Watertown, MA)

SUMMARY:
Body temperature measurement is one of the standard vital sign measurements in newborn babies in order assess their health status. Temperatures are taken on a regular basis throughout the newborn's stay on the well-baby floor. A temperature that is elevated above the normal range for age or depressed below the normal range for age may be a sign of illness in a newborn. There are many methods that may be used to record this temperature. Traditionally, axillary (under the arm) and rectal (in the rectum) sites have been used. Recently, a new method of temperature measurement has become available. Temporal artery thermometers are a non-invasive method to measure the baby's temperature by means of a light that is shone on the forehead that can read your baby's temperature quickly. It is not clear whether this method is accurate in the newborn period.

The purpose of this study is to evaluate the accuracy of temporal artery temperature measurement. This will be achieved by observing the axillary measurement, rectal temperature measurement, and temporal artery temperature measurement taken at approximately the same time in each infant. These measurements will be compared to each other to determine if temporal artery thermometry is as reliable a measurement as rectal and / or axillary temperature measurements.

We plan to compare

Hypothesis: Temporal artery thermometry of the immediate newborn infant is an accurate measurement of temperature in this age group.

ELIGIBILITY:
Inclusion Criteria:

* term newborns >/= 37 weeks gestational age
* late preterm infants >/= 35 weeks gestational age
* admitted to the well baby nursery following delivery
* < 24 hours of age

Exclusion Criteria:

* Infants < 35 weeks gestational age
* Infants currently under a radiant warmer or who have been under a radiant warmer < 1 hour prior to temperature measurement.

Max Age: 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2008-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Accuracy of temporal artery temperature compared to rectal and axillary temperature measurements. | All temperatures will be taken within 5 minutes of each other

CONTACTS AND LOCATIONS:
Overall Officials: Michael F. Bruno, MD, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Care Health Systems, Newark, Delaware, United States